CLINICAL TRIAL: NCT05918978
Title: Open-Label Extension Study to Evaluate the Long-term Safety and Efficacy of Efgartigimod in Adult Patients With Post-COVID-19 Postural Orthostatic Tachycardia Syndrome (PC-POTS) Who Completed Study ARGX-113-2104
Brief Title: Open Label Extension of Efgartigimod in Adults With Post-COVID-19 POTS
Acronym: POTS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the phase 2 results of the main study (ARGX-113-2104) showing that efgartigimod-treated PC-POTS patients had no clinically meaningful improvement, the decision has been made to terminate this open-label extension study (ARGX-113-2105) study.
Sponsor: argenx (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-113-2105
Record Dates: First submitted 2023-06-22; First posted 2023-06-26 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Post-COVID Postural Orthostatic Tachycardia Syndrome Postural Orthostatic Tachycardia Syndrome
Keywords: Tachycardia Post-COVID; Postural Orthostatic Tachycardia Syndrome efgartigimod
MeSH Terms: interventions — efgartigimod alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Efgartigimod (Experimental): Receive efgartigimod IV 10mg/kg infusions during a treatment period of 48 weeks
  Interventions: Drug: Efgartigimod

INTERVENTIONS:
Drug: Efgartigimod — Participants will receive efgartigimod IV 10 mg/kg open label, respectively.

SUMMARY:
The OLE study aims to investigate the safety, efficacy, pharmacodynamics (PD), pharmacokinetics (PK), and immunogenicity of efgartigimod in participants with post-COVID-19 postural orthostatic.

DETAILED DESCRIPTION:
Study ARGX-113-2105 is a long-term, single-arm, open-label, multicenter extension of the ARGX-113-2104 study, designed to evaluate the long-term safety of efgartigimod IV in adult patients with PC-POTS. Participants will be enrolled from both active and placebo arms of the ARGX-113-2104 study and will receive efgartigimod IV 10 mg/kg in the extension study without knowledge of their prior treatment arm. To be eligible to enroll in this study, participants must have completed the 24-week treatment period of the ARGX-113-2104 study and must not have permanently discontinued the IMP in that study.

ELIGIBILITY:
Inclusion Criteria:

1. The participant has completed the ARGX-113-2104 study without permanent discontinuation of IMP and agrees to directly roll over into the extension study without discontinuation of IMP.
2. The participant signs the informed consent form, and can comply with OLE study (ARGX-113-2105) protocol requirements.
3. The participant agrees to use contraceptives consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Contraceptive requirements are provided.
4. Female participants of childbearing potential must have a negative urine pregnancy test at baseline before receiving IMP.

Exclusion Criteria:

1. The participant has a clinically significant condition, based on the judgement of the Study Investigator, eg, laboratory abnormalities, 12-lead ECG readings, concomitant medical disease(s), etc., which may place them at undue risk or confound interpretation of study data.
2. The participant intends to become pregnant or start breastfeeding during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - UC Sand Diego Sulpizio Cardiovascular Center, La Jolla, California
  - Standford Movement Disorder Center, Palo Alto, California
  - North Shore University HealthSystem, Glenview, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University Hospitals, Neurology Clinical Trials, Cleveland, Ohio
  - Apex Trials Group, Fort Worth, Texas
  - Pioneer Clinical Research, Rosharon, Texas
  - Metrodora Institute, West Valley City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open-label study was an extension of ARGX-113-2104 study (NCT05633407) and was conducted at 9 sites in the United States from 26-Jun-23 to 15-Aug-24 in participants with post-coronavirus disease 2019 (COVID-19) postural orthostatic tachycardia syndrome (PC-POTS).
Pre-assignment Details: A total of 33 participants were rolled over from both active (efgartigimod) and placebo arms of the parent study ARGX-113-2104 (NCT05633407) to receive efgartigimod in this study. This study was terminated not for safety concerns but because the parent study found that efgartigimod intravenous (IV) provided no efficacy benefit in adult participants with PC-POTS.
Groups:
- Efgartigimod-Efgartigimod: Participants who received efgartigimod in parent study continued to receive efgartigimod 10 milligram/kilogram (mg/kg) via IV infusion from Day 1 once a week for the first 4 weeks (induction dosing period) and then once every 2 weeks for 42 weeks (maintenance dosing period).
- Placebo-Efgartigimod: Participants who received placebo in parent study received efgartigimod 10 mg/kg via IV infusion from Day 1 once a week for the first 4 weeks (induction dosing period) and then once every 2 weeks for 42 weeks (maintenance dosing period).
Period: Overall Study
Arm/Group | Efgartigimod-Efgartigimod | Placebo-Efgartigimod
Started | 20 | 13
Completed | 1 | 0
Not Completed | 19 | 13
Not completed — Study Terminated by Sponsor | 17 | 11
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on full analysis set (FAS) which included all enrolled participants.
Groups:
- Efgartigimod-Efgartigimod: Participants who received efgartigimod in parent study continued to receive efgartigimod 10 mg/kg via IV infusion from Day 1 once a week for the first 4 weeks (induction dosing period) and then once every 2 weeks for 42 weeks (maintenance dosing period).
- Total: Total of all reporting groups
Arm/Group | Efgartigimod-Efgartigimod | Placebo-Efgartigimod | Total
Number analyzed (Participants) | 20 | 13 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (11.38) | 38.0 (11.40) | 35.1 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 5 | 2 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 16 | 13 | 29
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 18 | 10 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With TEAEs, TESAEs and TEAESIs
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug. A serious adverse event (SAE) was any untoward medical occurrence that at any dose resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or any other medically important event. An adverse event of special interest (AESI) was an AE of scientific and medical concern specific to the sponsor's product or program. Treatment-emergent adverse events (TEAEs) were defined as AEs with onset on or after the first administration of study drug up to and including 60 days after the last study drug administration.
Time Frame: From the first dose of study drug (Day 1) up to 60 days post last dose of study drug, up to 383 days
Population: The safety analysis set (SAF) included all enrolled participants exposed to study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod-Efgartigimod | Placebo-Efgartigimod
Number analyzed (Participants) | 20 | 13
Participants
  TEAEs | 13 | 12
  TESAEs | 0 | 0
  TEAESIs | 7 | 5

2. Secondary Outcome: Change From Baseline to Weeks 24 and 48 in the COMPASS 31 (2-week Recall Version)
Description: Composite Autonomic Symptom Score (COMPASS) 31 modified version (2-week recall) is a self-rated questionnaire to evaluate the severity and distribution of autonomic symptoms in various autonomic nerve disorders. It consists of 31 questions in 6 weighted domains (orthostatic intolerance, vasomotor, secretomotor, gastrointestinal {GI}-mixed upper and diarrhea, bladder, and pupillomotor). A weighted total score of 0 (mild) to 100 (severe) was determined by adding a maximum raw score for each domain. Higher scores indicated a more severe degree of autonomic symptoms.
Time Frame: Baseline (Day 1) and Weeks 24 and 48
Population: The FAS included all enrolled participants. Only those participants with data collected at Baseline, Weeks 24 and 48 are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Efgartigimod-Efgartigimod | Placebo-Efgartigimod
Number analyzed (Participants) | 10 | 7
score on a scale
  Week 24 | 13.608 (29.7026) | 8.447 (18.1170)
  Week 48: number analyzed (Participants) | 1 | 0
  Week 48 | 1.780 |

3. Secondary Outcome: Change From Baseline to Weeks 24 and 48 in the MaPS
Description: The Malmö POTS Symptom Score (MaPS) score is a dedicated POTS symptom scoring questionnaire. The score consists of 12 questions that assess symptom burden related (tachycardia, palpitations, dizziness, presyncope) and unrelated to orthostatic intolerance (GI symptoms, insomnia, concentration difficulties). Participants graded their symptoms for the past 7 days using a numerical rating scale ranging from 0 (no symptoms) to 10 (very pronounced symptoms). The total score was calculated by summing up the items/individual items and range was 0 to 120 points, with higher scores indicating more severe symptoms.
Time Frame: Baseline (Day 1) and Weeks 24 and 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Efgartigimod-Efgartigimod | Placebo-Efgartigimod
Number analyzed (Participants) | 8 | 6
score on a scale
  Week 24 | -0.8 (22.02) | 10.3 (24.95)
  Week 48: number analyzed (Participants) | 1 | 0
  Week 48 | -17.0 |

4. Secondary Outcome: Percentage of Participants With Improved PGI-S at Weeks 24 and 48
Description: The Patient Global Impression-Severity (PGI-S) is a participant-rated, single-item scale to assess the severity of a health condition. The scale was used to assess the severity of symptoms over the past week (1-week recall) and overall experience of symptoms over the past 2 weeks (2-week recall). Both were rated on a 4-point type Likert scale, with scores ranging from 1 (none), 2 (mild), 3 (moderate), and 4 (severe). Higher scores indicate greater symptom severity. An "improved PGI-S" was defined by a change from baseline of -3, -2 and -1.
Time Frame: Baseline (Day 1) and Weeks 24 and 48
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Efgartigimod-Efgartigimod | Placebo-Efgartigimod
Number analyzed (Participants) | 8 | 5
percentage of participants
  Week 24, 1-week recall | 12.5 | 0
  Week 24, 2-week recall | 12.5 | 0
  Week 48, 1-week recall: number analyzed (Participants) | 4 | 4
  Week 48, 1-week recall | 25.0 | 0
  Week 48, 2-week recall: number analyzed (Participants) | 4 | 4
  Week 48, 2-week recall | 25.0 | 0

5. Secondary Outcome: Percentage of Participants With Improved PGI-C at Weeks 24 and 48
Description: The Patient Global Impression-Change (PGIC) is a single-item scale to capture the participant's perception of an overall change in their symptoms from start of study drug. It was rated on a 7-point Likert scale, with scores ranging from 1 (much better), 2 (somewhat better), 3 (a little better), 4 (no change), 5 (a little worse), 6 (somewhat worse), and 7 (much worse). Higher PGI-C scores signify worse outcome. An "improved PGI-C" was defined by a change from baseline of 1, 2 and 3.
Time Frame: Baseline (Day 1) and Weeks 24 and 48
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Efgartigimod-Efgartigimod | Placebo-Efgartigimod
Number analyzed (Participants) | 8 | 5
percentage of participants
  Week 24 | 100.0 | 100.0
  Week 48: number analyzed (Participants) | 4 | 4
  Week 48 | 100.0 | 75.0

6. Secondary Outcome: Change From Baseline to Weeks 24 and 48 in the PROMIS Fatigue Short Form 8a
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form 8a assesses the impact and perceived fatigue during the last 7 days. This validated 8-question scale has 5 response options, with scores ranging from 1 (not at all) to 5 (very much). Total scores ranged from 8 to 40; higher scores indicated higher fatigue levels and were converted to a T-score with a mean of 50 and standard deviation of 10. A decrease in T-score (negative change from baseline) indicated improvement in fatigue.
Time Frame: Baseline (Day 1) and Weeks 24 and 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Efgartigimod-Efgartigimod | Placebo-Efgartigimod
Number analyzed (Participants) | 8 | 5
T-score
  Week 24 | 3.0 (4.93) | 2.6 (9.74)
  Week 48: number analyzed (Participants) | 4 | 4
  Week 48 | -3.5 (3.42) | 1.0 (5.94)

7. Secondary Outcome: Change From Baseline to Weeks 24 and 48 in the PROMIS Cognitive Function Short Form 6a
Description: PROMIS Cognitive Function Short Form 6a assesses the frequency of cognitive difficulties experienced in the past 7 days. The questionnaire comprises 6 questions on subjective cognitive difficulties regarding a participant's concentration, memory, language, mental acuity, and perceived changes in cognitive functioning. The participant marks their response on a 5-point Likert scale (1: never and 5: very often). Scores ranged from 6 to 30; higher scores indicated worse perceived cognitive functioning and were converted to a T-score with a mean of 50 and standard deviation of 10. An increase in T-score (positive change from baseline) indicated better cognitive function.
Time Frame: Baseline (Day 1) and Weeks 24 and 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Efgartigimod-Efgartigimod | Placebo-Efgartigimod
Number analyzed (Participants) | 10 | 7
T-score
  Week 24 | -2.2 (7.36) | -4.0 (5.97)
  Week 48: number analyzed (Participants) | 1 | 0
  Week 48 | -8.0 |

8. Secondary Outcome: Percent Change From Baseline in Total IgG Levels at Weeks 24 and 48
Description: Blood samples for immunoglobulin G (IgG) analysis were collected at specified time points. Total IgG concentrations were quantified using validated methods at a central laboratory.
Time Frame: Baseline (Day 1) and Weeks 24 and 48
Population: The SAF included all enrolled participants exposed to study drug. Only those participants with data collected at Baseline, Weeks 24 and 48 are reported.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Efgartigimod-Efgartigimod | Placebo-Efgartigimod
Number analyzed (Participants) | 8 | 4
percent change
  Week 24 | 32.684 (28.6347) | -59.636 (6.2440)
  Week 48: number analyzed (Participants) | 1 | 0
  Week 48 | -10.360 |

9. Secondary Outcome: Serum Concentration of Efgartigimod
Description: Serum samples were collected at specified timepoints to determine the concentration of efgartigimod.
Time Frame: Pre-dose at Baseline (Day 1) and Weeks 1, 4, 12 and 24
Population: The pharmacokinetic analysis set (PKAS) included all enrolled participants who received at least 1 dose of efgartigimod and had at least 1 measured concentration of efgartigimod at a scheduled PK time point after start of dosing without protocol violations or events with potential to affect the PK concentration. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: microgram/milliliter (mcg/mL)
Arm/Group | Efgartigimod-Efgartigimod | Placebo-Efgartigimod
Number analyzed (Participants) | 18 | 9
microgram/milliliter (mcg/mL)
  Day 1: number analyzed (Participants) | 18 | 0
  Day 1 | 9 (4) |
  Week 1: number analyzed (Participants) | 16 | 8
  Week 1 | 10 (4) | 11 (4)
  Week 4: number analyzed (Participants) | 14 | 8
  Week 4 | 11 (4) | 12 (4)
  Week 12: number analyzed (Participants) | 8 | 9
  Week 12 | 3 (3) | 7 (6)
  Week 24: number analyzed (Participants) | 7 | 3
  Week 24 | 5 (5) | 2 (2)

10. Secondary Outcome: Number of Participants With ADAs Against Efgartigimod
Description: Blood samples were collected at specified timepoints to assess anti-drug antibodies (ADAs) against efgartigimod. ADA incidence reported here was defined as total number of participants with treatment-induced and treatment-boosted ADA. Treatment-induced ADA was defined as a baseline negative sample and at least 1 positive post-baseline sample. Treatment-boosted ADA was defined as a baseline positive sample and the titer value increased 4-fold or more compared to baseline.
Time Frame: From the first dose of study drug (Day 1) up to Week 48
Population: The SAF included all enrolled participants exposed to study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod-Efgartigimod | Placebo-Efgartigimod
Number analyzed (Participants) | 20 | 13
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: From the first dose of study drug (Day 1) up to 60 days post last dose of study drug, up to 383 days
Description: Analysis was performed on the SAF. Laboratory abnormalities were reported as AEs.
Arm/Group | Efgartigimod-Efgartigimod | Placebo-Efgartigimod
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/13
Other Adverse Events (participants affected / at risk) | 13/20 | 12/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efgartigimod-Efgartigimod (N=20) | Placebo-Efgartigimod (N=13)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (5) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (3) | 0 (0)
Energy increased (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 3 (6)
Injection site bruising (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Contrast media reaction (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 5 (5) | 1 (1)
Gastrointestinal bacterial overgrowth (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time shortened (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (2) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (3)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Migraine (Nervous system disorders) | 1 (2) | 1 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin tightness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vasodilatation (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated not for safety concerns but because the parent study found that efgartigimod IV provided no efficacy benefit in adult participants with PC-POTS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/78/NCT05918978/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT05918978/SAP_001.pdf